CLINICAL TRIAL: NCT00417781
Title: A Follow-up, Family Study on Attention-deficit Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: 9361700470; NHRI-EX94-9407PC (Other: National Health Research Institute); NHRI-EX95-9407PC (Other: National Health Research Institute); NHRI-EX96-9607PC (Other: National Health Research Institute); NHRI-EX97-9707PC (Other: National Health Research Institute); NHRI-EX98-9507PC (Other: National Health Research Institute)
Record Dates: First submitted 2006-12-31; First posted 2007-01-04 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD, adolescence, family study, endophenotype, outcome
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: Attention deficit hyperactivity disorder (ADHD), characterized by inattention, hyperactivity and impulsivity, is an early onset, common (5-10% worldwide; 7.5% in Taiwan), clinically heterogeneous, impairing disorder. Despite the abundance of research on ADHD, the vast majority of samples have been limited to Caucasians; there is limited information about the expressions, patterns, correlates, and outcomes for ADHD in the Taiwanese population.

Specific Aims:

1. to investigate the neuropsychological functioning, and psychiatric, academic, and social outcomes of ADHD at adolescence;
2. to examine the psychopathology and neuropsychological functioning among parents and siblings of ADHD probands;
3. to determine the components of ADHD and neuropsychological functioning with the greatest familial recurrence risks; and
4. to validate the classification of ADHD and comorbid subtypes of ADHD using psychosocial, familial, neuropsychological and longitudinal data.

Subjects and Methods: This 5-year proposal consists of two parts: (1) a 3 year-retrospective cohort study and family study design; and (2) a 2 year-prospective cohort study design. Several Chinese version of rating scales will be prepared in the first 6 months. The sample will consist of probands with (n=180) and without (n=90) ADHD, ages 11-16, recruited from the Children's Mental Health Center, NTUH and an epidemiological study. The ADHD diagnosis has been made 3-6 years ago prior to recruitment. Probands and their parents will be assessed using the following measures (n=810) in the first 3 years. Only probands will be reassessed in the last 2 years. The measures will include a psychiatric interview using K-SADS-E and self-reports covering the individual and familial/environmental domains; and neuropsychological tests (WISC-III, CPT, WCST, CANTAB). The informants include probands and their parents and teachers.

Long-term Objectives: The long-term objectives are to identify the endophenotypes that are close to the biological expression of genes underlying ADHD, to determine the familial aggregation and its specificity regarding the components of ADHD, and neuropsychological deficit, and to identify the impact of ADHD on academic, psychiatric, family, and social outcomes; and to identify a cohort of families with ADHD for future neuroimaging, neurophysiological, and molecular genetic studies.

DETAILED DESCRIPTION:
(A) Specific Aims

The ultimate goals of this family study are to identify the endophenotypes that are closer to the biological expression of genes underlying ADHD, to identify patterns of familial aggregation with regards to ADHD and neuropsychological function, to examine the impact of ADHD on family functioning and parental psychosocial adjustment, and to characterize the long-term outcome of ADHD at adolescence in a Taiwanese sample. We propose to replicate previous studies on ADHD using a novel approach (an ambispective follow-up, bottom-up family study design using a mixed clinical and epidemiological sample) to validate the findings of previous studies in terms of the correlates, patterns, expression, outcome, and familial aggregation for ADHD and to attempt to determine whether neurological, and neuropsychological dysfunctioning also run in ADHD probands. With the accomplishment of these goals, this study will resolve controversies over inconsistent findings in previous studies and contribute to the literature on the validity of ADHD and ADHD comorbid subtypes using family data. The specific aims of this study are:

1. Follow-up component:

   1. to explore the potential risk factors for the developing ADHD;
   2. to investigate the expression and patterns of ADHD at adolescence in terms of symptoms, neuropsychological, neurological, familial, school and social functions;
   3. to examine the symptoms continuity and the determinants of persistent ADHD symptoms;
   4. to identify the symptomatic, academic, and social outcomes of ADHD at early and late adolescence, including the use of tobacco, betel nut, alcohol and drug; and
   5. to validate the comorbid subtypes of ADHD using psychopathological, neuropsychological, behavioral, familial and social correlates.
2. Family study component:

   1. to examine the psychopathology and neuropsychological functioning among parents and probably siblings of ADHD probands in comparison with those of control probands; and
   2. to identify the most familial correlated components of ADHD symptoms and neuropsychological measures.

A. Specific Hypotheses

The major research questions for the current proposal generated from prior research by our group and others are listed below. Under each question, specific hypotheses are provided:

1. What are the major adolescent and young adult outcomes for children with ADHD? (Outcome of ADHD)

   1. Children with ADHD will be more likely to have comorbid psychiatric disorders such as oppositional defiant disorder, conduct disorder, depression, and substance use such as initial use of nicotine, betel nut, and alcohol at adolescence and depression, substance abuse, and antisocial personality disorder at young adulthood.
   2. Academic underachievement, impaired functioning in several social domains, interpersonal difficulties, and low self-esteem will be apparent at adolescence and young adulthood.
2. What are the correlates and endophenotype of ADHD? (Validity of ADHD)

   a. Adolescents with ADHD will have more prenatal exposure to alcohol and nicotine, family dysfunction, parent-child conflict, sleep-related problems, somatic complaints, and neurological and neuropsychological dysfunctioning than those without ADHD.
3. What are the specific components of ADHD that are familial?

   1. We hypothesize that parents of children with ADHD are at higher risks for ADHD and inattention will demonstrate more apparent family aggregation than hyperactivity.
   2. We also anticipate that deficit in executive function such as impaired working memory, impulsivity, and problem-solving difficulties will be familial among individuals with ADHD.
   3. In addition, associations between risk factors, and correlates that have not been addressed previously are also investigated post hoc. These analyses will be corrected for multiple comparisons.

Significance and Background (deleted here) (E) Research Design and Methods This is a 5-year project with the first three years of a retrospective cohort study and family study designs and the last two years of a prospective follow-up cohort study design.

A.1: The First Three-Year Study (2005.1~2007.12):

The major tasks of the first 3-year of this study consisted of three parts: (1) 6 months-development of several rating scales for adolescent and adult subjects, K-SADS-E interview training, pilot study of the Cambridge Neuropsychological Test Automated Batteries, and recruitment of subjects; (2) 2 years and 3 months-completion of recruitment and assessments of 180 ADHD families and 90 control families (n=810); and (3) 3 months-data management and analyses for the adolescent outcome and family aggregation of these 270 families and preparation for the follow-up study in the young adulthood.

A.1.1: Preparation phase-the first 6 months (2005.1~2005.6)

1. Reliability and validity of instruments The Chinese version of the Conners Parent Rating Scale-Revised Short Form (CPRS-R: S), Conners Teacher Rating Scale-Revised Short Form (CTRS-R: S), Adult ADHD rating scale (ASRS), and Adult Self-Report Inventory (ASRI) will be prepared with culture-relevant colloquial expressions by the experienced child psychiatrists and professional translators.
2. K-SADS-E and SAICA semi-structural interview training The interviewers will be trained to conduct the K-SADS-E interviews for parent report on themselves and probands, and proband report on themselves by the PI and staff child psychiatrists. (The details of training courses will be provided upon request).
3. Training for administration and pilot study of neuropsychological tests including the Cambridge Neuropsychological Test Automated Batteries (CANTAB), CPT, and WSCT.

A.1.2: Follow-up Studies for Children with ADHD-2 years and 3 months (2005.7~2007.9)

a. Description of Subjects

1. 1: Selection of Subjects The sample will consist of two groups: one exposed group including aged 12 to 15 adolescents with ADHD and one unexposed group including adolescents without ADHD. Their parents will be recruited in the family study. Their psychiatric diagnoses were made 3-6 years ago either at a clinical setting or in an epidemiological study. Recruitment will stop when we will have approximately 180 probands with ADHD and 90 control probands.

   1. Inclusion Criteria The inclusion criteria for the exposed group are (1) that subjects either had the clinical diagnosis of DSM-IV ADHD, which was made by a full-time child psychiatrist at the first visit and following visits or by a child psychiatrist using the K-SADS-E as the second-stage case ascertainment at an epidemiological study; (2) the diagnoses of ADHD were made 3-6 years ago; (3) their ages range from 12 to 15 when we conduct study; (4) subjects have at least one sibling aged 6-18 and live with at least one biological parent; and (5) subjects and their family consent to participate in this study.

      The inclusion criteria for the unexposed group are (1) that subjects were assessed either at a clinical setting or in an epidemiological study same as to those in the exposed group 6 years ago; (2) their ages range from 12 to 15 when we conduct study; (3) subjects have at least one sibling aged 6-18 and live with at least one biological parent; and (4) subjects and their family consent to participate in this study.
   2. Exclusion Criteria The subjects, including those who in the exposed and unexposed groups, will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, Organic Psychosis, Mental Retardation, or Pervasive Developmental Disorder. Moreover, the subjects will be excluded from the unexposed group if have a history of the following condition as defined by DSM-IV: ADHD, ODD, or CD in addition to the above exclusion criteria. a.2: Source of Subjects Half of the subjects will be recruited from the Department of Psychiatry, National Taiwan University Hospital and half from the community in Taipei city based on the diagnoses in a epidemiology survey for ADHD.
2. Procedures A letter and telephone contact with explanation of the purpose and procedure of this study and reassurance of confidentiality will be done before the recruitment of subjects, followed by face-to-face explanation and written informed consent. The subjects and their parents will be interviewed separately to provide information about the subjects' family composition, prenatal, developmental, and medical history, psychiatric diagnoses, and social functioning. CANTAB and other neuropsychological tests will be administered to probands and their parents. We will implement a quality control procedure consisting of verification of the interviews of 20% of the sample. These subjects will have their interview verified with audiotape, which will be reviewed by a blinded rater. The child and parent self-reported questionnaires will be administered either before or after child and parent interviews. We will interview 270 families (# N of assessments = 810). For the second-part of follow-up study at late adolescence (2008.1~2009.9), we will try to obtain corresponding information such as the addresses, telephone numbers, and email addresses of their relatives or friends close to them in order to decrease the loss of follow-up rates.

A.1.3: Data Analysis and Manuscript Preparation for the first part of study-Adolescent Outcome (2007.10~2007.12) The research team will concentrate on data management and analysis of the information gathered in the first three years to understand the adolescent outcome and endophenotype of ADHD. We will also try to prepare several manuscripts for publication.

A.3: Interviews and Psychiatric Diagnosis: Interviewers will be supervised by staff child psychiatrists. We developed a formal training package including an overview of the study and its methods, the diagnostic instruments, and detailed descriptions of the instruments and interview procedures. DVD of psychiatric interviews with adolescents and adults with ADHD and other major diagnostic categories are available for training and developing inter-rater reliability. The quality control of interview will be carried out continuously.

The PI got her training in best estimate for diagnoses in her doctoral study at Yale. The best estimate diagnosis, based upon all available information (interviews, questionnaires, family histories, and medical records), will be made by the PI who will be blind to the diagnostic status of the proband and who will not be involved in direct interviews of any of the probands or parents.

B. Measures B.1: Interviews for Psychiatric Diagnostic Information and Social functioning using the Chinese K-SADS-E for making diagnosis of probands and their siblings and parents; and the Social Adjustment Inventory for Children and Adolescents B.1.2: Self-reported measures The assessments will cover individual and familial/environmental vulnerability factors. They include measures of symptomatology, temperament/personality, psychopathology, competence, pubertal status, sleep patterns as well as familial and school functioning (Table 1). Chinese versions of these self-reported scales will be available including CBCL, CTRS-R:S, CPRS-R:S, EPQ-JR, PDS, MES, DOTS, SAICA-C, PBI-C, FACS-C, ASRI, and DAS.

Long-term Objectives: The long-term objectives are to identify the endophenotypes that are close to the biological expression of genes underlying ADHD, to determine the familial aggregation and its specificity regarding the components of ADHD, and neuropsychological deficit, and to identify the impact of ADHD on academic, psychiatric, family, and social outcomes; and to identify a cohort of families with ADHD for future neuroimaging, neurophysiological, and molecular genetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Community-based sample for the development of several Chinese versions of instruments: SNAP-IV, SDQ, ASRI, and ASRS.
* ADHD follow-up family studies (ADHD group): (1) that subjects either had the clinical diagnosis of DSM-IV ADHD, which was made by a full-time child psychiatrist at the first visit and following visits or by a child psychiatrist using the K-SADS-E as the second-stage case ascertainment at an epidemiological study; (2) the diagnoses of ADHD were made 3-6 years ago; (3) their ages range from 12 to 15 when we conduct study; (4) subjects have at least one sibling aged 6-18 and live with at least one biological parent; and (5) subjects and their family consent to participate in this study.
* (control group)(1) that subjects were assessed either at a clinical setting or in an epidemiological study same as to those in the exposed group 6 years ago; (2) their ages range from 12 to 15 when we conduct study; (3) subjects have at least one sibling aged 6-18 and live with at least one biological parent; and (4) subjects and their family consent to participate in this study.

Exclusion Criteria:

* The subjects, including those who in the exposed and unexposed groups, will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, Organic Psychosis, Mental Retardation, or Pervasive Developmental Disorder. Moreover, the subjects will be excluded from the unexposed group if have a history of the following condition as defined by DSM-IV: ADHD, ODD, or CD in addition to the above exclusion criteria.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Community-based sample & children with ADHD and their families
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2005-01; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chiang HL, Gau SS. Impact of executive functions on school and peer functions in youths with ADHD. Res Dev Disabil. 2014 May;35(5):963-72. doi: 10.1016/j.ridd.2014.02.010. Epub 2014 Mar 11. PMID 24636025
- [Derived] Gau SS, Chiang HL. Association between early attention-deficit/hyperactivity symptoms and current verbal and visuo-spatial short-term memory. Res Dev Disabil. 2013 Jan;34(1):710-20. doi: 10.1016/j.ridd.2012.10.005. Epub 2012 Nov 5. PMID 23137723
- [Derived] Wu SY, Gau SS. Correlates for academic performance and school functioning among youths with and without persistent attention-deficit/hyperactivity disorder. Res Dev Disabil. 2013 Jan;34(1):505-15. doi: 10.1016/j.ridd.2012.09.004. Epub 2012 Oct 11. PMID 23063730
- [Derived] Gau SS, Lin YJ, Cheng AT, Chiu YN, Tsai WC, Soong WT. Psychopathology and symptom remission at adolescence among children with attention-deficit-hyperactivity disorder. Aust N Z J Psychiatry. 2010 Apr;44(4):323-32. doi: 10.3109/00048670903487233. PMID 20307165